CLINICAL TRIAL: NCT00125762
Title: Comparison of FibroScan With Histological Evaluations of Liver Fibrosis in Patients With Hepatitis B and C Presenting for Liver Biopsy
Brief Title: FibroScan in Patients With Hepatitis B and C Presenting for Liver Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afdhal, Nezam, M.D. (Individual)
Collaborators: Echosens (Industry)
Responsible Party: Principal Investigator, Nezam H. Afdhal, Professor of Medicine, Part-time, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004P000251
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Cirrhosis; Hepatitis B; Hepatitis C
MeSH Terms: conditions — Fibrosis; Hepatitis B; Hepatitis C

STUDY DESIGN:
Masking Description: Investigator unaware of biopsy results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm undergoing FibroScan (Experimental): Single arm active comparison of biopsy to vibration controlled elastography
  Interventions: Device: FibroScan

INTERVENTIONS:
Device: FibroScan

SUMMARY:
This study will examine the effectiveness of the FibroScan device in differentiating fibrosis in patients with hepatitis B and C. The FibroScan measures liver stiffness and will be correlated to the liver biopsy to see if it can diagnose the stage of liver disease. Patients who are scheduled to have a liver biopsy will also have a fibroscan and the stiffness will be correlated with the biopsy stage.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Co -Primary Aims:

* Diagnosis of cirrhosis in patients with chronic viral hepatitis B and C;
* Correlation of the FibroScan measurement with Metavir liver fibrosis scores by differentiating no/mild fibrosis (F0-F1) from severe fibrosis (F2-F4).

STUDY DESIGN:

This is a multi-center study in which the FibroScan measurements will be collected prospectively from patients with chronic hepatitis B and C virus presenting for liver biopsy. The study duration will be 12 months. The study will initially have 3 investigational sites in the United States. Up to 3 more investigational sites may be identified to participate in the trial.

Study Sites:

Initially the following three sites will participate in the trial:

Duke University Medical Center, Durham, NC: Keyur Patel, M.D.; Beth Israel Deaconess Medical Center and Harvard Medical School, Boston, MA: Nezam H. Afdhal, M.D.; St. Louis University, St. Louis, MO: Bruce R. Bacon M.D.

Study Population:

Subjects with chronic liver diseases secondary to chronic hepatitis C and hepatitis B, undergoing a liver biopsy as the standard of care for their disease, will be eligible for the study. Subjects with hepatitis C, co-infected with other infectious viral diseases, such as hepatitis B or HIV-1, or both, may also be candidates for study enrollment provided the inclusion/exclusion criteria are met.

The subjects must be scheduled for liver biopsy either prior to treatment (treatment naïve) or, if previously treated, they must have been off treatment for at least three (3) months. The time between the date of the FibroScan reading and the date of biopsy must not exceed six (6) months.

Sample Size:

A total of at least 300 evaluable patients (males and females) will be enrolled in this study. Enrollment will be considered competitive with no site enrolling more than 50% of the study population. Sample size is based on a prevalence of 20% cirrhosis.

Subject Inclusion Criteria:

* Subject is able to give informed consent for this study and agrees to provide a blood sample.
* Subject must be at least 18 years of age.
* Subject has had or will have a liver biopsy for chronic liver disease, secondary to HBV or HCV or within 6 months of FibroScan (experimental cohort 1 only).
* Subjects who have hepatitis C (HCV) or hepatitis B (HBV) should be treatment naïve or off interferon therapy or nucleoside/nucleotide analogs for HBV for a minimum of 3 months prior to the FibroScan and liver biopsy.

Subject Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Confirmed diagnosis and/or history of malignancy, or other terminal disease.
* Uninterpretable biopsy specimen.
* Missing critical clinical, biochemical and/or demographic information.
* Receiving anti-viral therapy for infection of HCV or HBV within 3 months prior to the FibroScan and liver biopsy.
* Subject with other chronic liver disease, including Wilson's disease, alpha 1-antitrypsin deficiency, cholestatic liver disease, or hemochromatosis.
* Patient with clinical ascites
* Patients with morbid obesity defined as a body mass index (BMI) of greater than or equal to 40.
* Patients who are pregnant
* Patients who have an implantable cardiac device such as defibrillator or pacemaker

SAMPLE REQUIREMENTS and TESTING:

A minimum of 8 valid measurements will be obtained for each subject from the right lobe of the liver. The tip of the probe transducer will be covered with coupling gel and placed on the skin, between the ribs at the level of the right lobe of the liver. The operator, assisted by an ultrasonic time motion image, will locate a portion of the liver that is at least 4cm thick and free of large vascular structures. The depth of measurement will be between 25 mm and 65 mm. During the acquisition subjects will lie on their back with the right arm behind the head, in a similar position to that used for liver biopsy. The physician will take the measurements with the probe placed in the intercostal space. The median value of the estimates will be kept as the elasticity value of the liver for a given patient. The entire examination should last approximately 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to give informed consent for this study and agrees to provide a blood sample.
* Subject must be at least 18 years of age.
* Subject has had or will have a liver biopsy for chronic liver disease, secondary to HBV or HCV or within 6 months of FibroScan (experimental cohort 1 only).
* Subjects who have hepatitis C (HCV) or hepatitis B (HBV) should be treatment naïve or off interferon therapy or nucleoside/nucleotide analogs for HBV for a minimum of 3 months prior to the FibroScan and liver biopsy.

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Confirmed diagnosis and/or history of malignancy, or other terminal disease.
* Uninterpretable biopsy specimen.
* Missing critical clinical, biochemical and/or demographic information.
* Receiving anti-viral therapy for infection of HCV or HBV within 3 months prior to the FibroScan and liver biopsy.
* Subject with other chronic liver disease, including Wilson's disease, alpha 1-antitrypsin deficiency, cholestatic liver disease, or hemochromatosis.
* Patient with clinical ascites.
* Patients with morbid obesity defined as a BMI of greater than or equal to 40.
* Patients who are pregnant.
* Patients who have an implantable cardiac device such as defibrillator or pacemaker.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2008-05-01 (Actual); Study Completion 2008-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nezam H Afdhal, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - BIDMC, Boston, Massachusetts
  - Bruce Bacon M.D., St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Afdhal NH, Bacon BR, Patel K, Lawitz EJ, Gordon SC, Nelson DR, Challies TL, Nasser I, Garg J, Wei LJ, McHutchison JG. Accuracy of fibroscan, compared with histology, in analysis of liver fibrosis in patients with hepatitis B or C: a United States multicenter study. Clin Gastroenterol Hepatol. 2015 Apr;13(4):772-9.e1-3. doi: 10.1016/j.cgh.2014.12.014. Epub 2014 Dec 18. PMID 25528010

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Arm: All patients received a liver biopsy and a FibroScan
Period: Overall Study
Arm/Group | Active Arm
Started | 907
Completed | 748
Not Completed | 159

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Undergoing FibroScan: Single arm active comparison of biopsy to vibration controlled elastography
  FibroScan
Arm/Group | Single Arm Undergoing FibroScan
Number analyzed (Participants) | 907
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 907
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis is for patients who completed both the liver biopsy and the FibroScan
  Participants
    number analyzed (Participants) | 748
    Female | 257
    Male | 491
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 586
  More than one race | 0
  Unknown or Not Reported | 321
Region of Enrollment [Number; unit: participants]
  United States | 907

OUTCOME MEASURES:

1. Primary Outcome: Diagnosis Performance of VCTE for Determination of Cirrhosis (Metavir F4) in Patients With Chronic Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV)
Description: VCTE was used to diagnose cirrhosis F4 in 748 patients undergoing liver biopsy and VCTE within a 28 day time period.
Time Frame: 28 days
Population: 748 patients were eligible for analysis with matching valid liver biopsies and VCTE measurements.
Measure: Mean (95% Confidence Interval); unit: ROC area
Arm/Group | Single Arm Undergoing FibroScan
Number analyzed (Participants) | 748
ROC area | 0.92 [0.87 to 0.95]

2. Primary Outcome: Diagnostic Accuracy of VCTE for the Prediction of Metavir Fibrosis Scores by Differentiating no/Mild (F0/F1) From Severe Fibrosis (F2 - F4)
Description: 95% CI for Metavir Fibrosis stage 0 -1 consistent with no or mild fibrosis compared to Metavir 2 - 4 which represents significant fibrosis or cirrhosis
Time Frame: Liver Biopsy and VCTE within a time frame of 6 months
Population: 456 patients with matching liver biopsy and fibroscan
Measure: Mean (95% Confidence Interval); unit: ROC area
Arm/Group | Single Arm Undergoing FibroScan
Number analyzed (Participants) | 456
ROC area | 0.89 [0.83 to 0.92]

ADVERSE EVENTS:
Time Frame: During FibroScan
Arm/Group | Active Arm
All-Cause Mortality (participants affected / at risk) | 0/907
Serious Adverse Events (participants affected / at risk) | 0/907
Other Adverse Events (participants affected / at risk) | 0/907

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No